CLINICAL TRIAL: NCT03321266
Title: A Retrospective Review of the Use of the Cook Biodesign® Fistula Plug (C-FPS-0.2, C-FPS-0.4, and C-FPS-0.7) to Treat Anorectal Fistulas
Brief Title: Retrospective Review of the Cook Biodesign® Fistula Plug to Treat Anorectal Fistulas
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 17-03
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Anorectal Fistula
Keywords: Fistula plug
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated for a anorectal fistula: Patients who were treated for a anorectal fistula with a Biodesign Fistula plug
  Interventions: Device: Cook Biodesign® Fistula Plug

INTERVENTIONS:
Device: Cook Biodesign® Fistula Plug — The Cook Biodesign® Fistula Plug is for implantation to reinforce soft tissue for repair of Anorectal fistulas.

SUMMARY:
The study is a retrospective review of the use of the Biodesign® Fistula Plug (C-FPS-[X]). A total of 73 patients will be enrolled who have had a fistula plug placed to treat anorectal fistulas and will therefore be eligible for statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had surgery to treat anorectal fistula where the Biodesign® Fistula Plug was placed during the procedure

Exclusion Criteria:

* Patients not receiving the Biodesign® Fistula Plug for treatment of their anorectal fistula

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients implanted with the Cook Biodesign Fistula Plug at each of the participating institutions through 31 Dec 2016 will be included in the retrospective data collection regardless of outcome. A patient must have at least one follow-up visit.
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Rate of fistula closure | up to 2 years
  Absence of drainage from the external fistula opening with complete epithelialization of the external fistula opening upon clinical exam.

CONTACTS AND LOCATIONS:
Overall Officials: Adal Saeed, MD, Principal Investigator — St Josef's Hospital, Wiesbaden
Locations (4):
- United States (3):
  - University of Louisville School of Medicine, Louisville, Kentucky
  - Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana
  - University Surgical Associates, Providence, Rhode Island
- St Josef's Hospital, Wiesbaden, Germany